CLINICAL TRIAL: NCT05786677
Title: Effect of Physiotherapy Protocol in Treatment of Depression: Longitudinal Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahitab Momen Gamal-Eldien Elansary, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mahitab_2023
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Fibromyalgia; Depression
MeSH Terms: conditions — Fibromyalgia; Depression | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with fibromyalgia and depression (1) (Experimental): Patients in this group will receive physiotherapy protocol and medications.
  Interventions: Other: Physiotherapy protocol; Drug: Selective serotonin reuptake inhibitors (SSRI)
- Patients with fibromyalgia and depression (2) (Active Comparator): Patients in this group will receive medications only.
  Interventions: Drug: Selective serotonin reuptake inhibitors (SSRI)
- Patients with depression only (1) (Experimental): Patients in this group will receive physiotherapy protocol and medications.
  Interventions: Other: Physiotherapy protocol; Drug: Selective serotonin reuptake inhibitors (SSRI)
- Patients with depression only (2) (Active Comparator): Patients in this group will receive medications only.
  Interventions: Drug: Selective serotonin reuptake inhibitors (SSRI)

INTERVENTIONS:
Other: Physiotherapy protocol — the physiotherapy protocol which will include: 4. Exercise in the form of: d. Breathing exercise e. Aerobic exercise (walking on treadmill with a speed of 3 miles per hour and 0% inclination) f. Bridging exercise 5. Manual techniques in the form of:
  1. Suboccipital release
  2. Diaphragm release
  3. Clavi-pectoral myofascial release 6. Home Routine
  c. Hot tub bath for 30 minutes d. Breathing exercise
  Arms: Patients with depression only (1); Patients with fibromyalgia and depression (1)
Drug: Selective serotonin reuptake inhibitors (SSRI) — Selective serotonin reuptake inhibitors (SSRIs)

SUMMARY:
The purpose of his study is to investigate the effect of physiotherapy protocol in management of depression in patients with fibromyalgia and in patients with psychogenic depression.

DETAILED DESCRIPTION:
This study will investigate the effect of physiotherapy protocol in management of depression in patients with fibromyalgia and in patients with psychogenic depression.

ELIGIBILITY:
Inclusion Criteria:

1. Fibromyalgia patients will be included if they meet the diagnosis of FM according to the American College Rheumatology (ACR), diagnosed with depression and referred by a physician.
2. Patients diagnosed with mild and moderate forms of major depression.
3. Their ages range from 20- 60 years old.
4. Patients willing and able to participate in a physiotherapy program and capable of doing physical exercise on their own.

Exclusion Criteria:

1. severe spinal injuries
2. severe musculoskeletal abnormalities
3. inflammatory rheumatic diseases
4. respiratory or cardiac pathologies
5. Any vestibular, visual or neurological dysfunction affecting balance.
6. History of suicidal attempts
7. Severe depression
8. Suffering from severe somatic or psychiatric disorders.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Assessing the change in severity of respondents' depression | at baseline, after 2 weeks of intervention, after 4 weeks of intervention and after one month and two months of end of treatment period
  Assessment will be done by using Arabic version of Beck Depression Inventory (BDI) which is designed to rate the severity of respondents' depression in the weeks preceding questionnaire completion. Each of the 21 questions presents four different statements and asks respondents to select the option that best represents them. Statements refer to depressive states in varying degrees of severity (from "I do not feel sad" to "I am so sad or unhappy that I can't stand it"), and this is reflected in the scoring process which assigns higher values to responses indicating more acute symptoms of depression. The total score can range from 0 to 63 points, with a total score of 0-9 points indicating minimal depression, 10-18 points mild, 19-29 points moderate, and 30-63 points severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Mahitab Momen, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic faculty of physica therapy cairo university, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided